CLINICAL TRIAL: NCT04397302
Title: Reverse Remodeling is Associated With Hemodynamic Improvement and Stabilization in Outpatients With Heart Failure With Reduced Ejection Fraction Treated With Sacubitril/Valsartan: an Echocardiographic Study
Brief Title: Role of Sacubitril/Valsartan in the Improvement of Heart Failure With Reduced Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Italian Society of Cardiology (Other)
Collaborators: Università degli Studi di Brescia (Other); Federico II University (Other); Ospedali Riuniti di Foggia (Other); University Of Perugia (Other); Monaldi Hospital (Other); University of Messina (Other); University of Siena (Other); University of Salerno (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Azienda Ospedaliero-Universitaria di Parma (Other); Azienda Unita Sanitaria Locale di Piacenza (Other)
Responsible Party: Principal Investigator, Frank Lloyd Dini, MD, Clinical Professor, Italian Society of Cardiology
Other Study IDs: 20190015213
Record Dates: First submitted 2020-05-04; First posted 2020-05-21 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure, Left Sided; Left Ventricular Dysfunction; Ventricular Remodeling
Keywords: Angiotensin-receptor neprilysin-inhibitor; Heart failure with reduced ejection fraction; Left ventricular filling pressure; Left ventricular reverse remodeling
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left; Ventricular Remodeling | interventions — Hemodynamics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 376 Days
Biospecimen Retention: Samples Without DNA — Serum, Plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Role of Sacubitril/Valsartan in Hemodynamic and Echocardiographic Improvement of Heart Failure With Reduced Ejection Fraction — Reverse Remodeling is Associated With Hemodynamic Improvement and Stabilization in Outpatients With Heart Failure With Reduced Ejection Fraction Treated With Sacubitril/Valsartan: an Echocardiographic Study

SUMMARY:
This prospective study evaluates the mechanisms of benefit of sacubitril/valsartan in a population of outpatients with heart failure with reduced ejection fraction, to investigate the relationship between the effects on left ventricular ejection fraction and volumes and noninvasively hemodynamic echo-derived parameters, as cardiac output and left ventricular filling pressure.

DETAILED DESCRIPTION:
Therapeutic interventions were made according to a titration protocol in stable optimal medical therapy. Therapy with sacubitril/valsartan was introduced after a 48-hour wash-out of an ACE inhibitor or after a 24-hour wash-out of an angiotensin receptor antagonist. Doses of sacubitril/valsartan were optimized to individual tolerability.

Echocardiography was performed at baseline and after 12 months. LV end-diastolic and end-systolic volumes were calculated according to the biplane Simpson's method according to the recommendations of the American Society of Echocardiography and European Association of Cardiovascular Imaging. Doppler examinations included assessment of early diastolic filling velocity and early diastolic mitral annular velocity, an averaged E/e' ≥ 13 was considered a surrogate marker of increased filling pressure.

The LV stroke volume was calculated as the product of the LV outflow tract area and the time-velocity integral of the aortic flow velocity or was evaluated as the difference between LVEDV and LVESV. The LVSV index was estimated as LVSV divided by body surface area. Cardiac output (CO) was measured as stroke volume times heart rate, and the cardiac index was estimated by dividing CO by body surface area.

Patients who presented reverse remodeling were considered those exhibiting a ≥ 10% increase in ejection fraction and ≥15% reduction in end-systolic volume compared to baseline.

The accuracy of the sources data was verified by using in-hospital medical records, computerized or paper, by checking data from ultrasound images, laboratory reports or ambulatory cardiological tests.

Detailed information on patients' medical history, including medications and loop diuretic doses, was recorded for each patient. Patients' functional status was determined according to the classification of the New York Heart Association. Creatinine, B-type natriuretic peptide and amino-terminal pro-type B-natriuretic peptide levels were measured using standard laboratory methods. The estimated glomerular filtration rate was calculated by the Modification of Diet in Renal Disease formula.

Patients were removed from therapy with sacubitril/valsartan or assessment for non-adherence to treatment or persistent drug-related adverse event with his/her willingness to discontinue treatment.

Continuous measures were expressed as the mean value ± SD or median and interquartile range (IRQ) for normally and non-normally distributed variables, respectively. Continuous data were compared using paired and independent samples Student t-test or ANOVA when appropriate. Categorical variables were presented as percentages and were compared using Chi-square or McNemar test. Mann-Whitney, Kruskal-Wallis and Wilcoxon tests were used to analyze non-normally distributed variables. All differences were considered significant at the p = 0.05 level. Data were analyzed with SPSS version 23.0 (IBM Corp., Armonk, NY).

ELIGIBILITY:
INCLUSION CRITERIA

* Ambulatory patients on stable optimal medical therapy
* History of HF and LVEF ≤ 40%
* II-III NYHA class

EXCLUSION CRITERIA

* History of congenital heart disease
* Severe valvular disease or valvular surgery
* Recent acute coronary syndromes or stroke
* Poor acoustic windows or missing data.
* Death or uncompleted follow-up evaluation
* Cardiac surgery interventions
* Cardiac resynchronization therapy
* Coronary or mitral interventions

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participants were recruited from a population of ambulatory patients with heart failure and reduced LV ejection fraction, being treated by Units of Cardiology in 12 Italian University hospitals.
Sampling Method: Probability Sample
Enrollment: 652 (Actual)
Dates: Start 2019-01-13 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Cardiac Output after 12 months of treatment | March, 16 th 2019 - March,16th 2020
  Cardiac Output (in L/min) is a variable measured by echocardiography as the product of LV stroke volume (in mL/beat) and heart rate (in bpm).

SECONDARY OUTCOMES:
Change from baseline in Left Ventricular Filling Pressure after 12 months of treatment | March, 16th 2019 - March,16th 2020
  Left ventricular filling pressure is calculated by Doppler Echocardiography as the ratio of early diastolic filling velocity (E wave, m/s) and early diastolic mitral annular velocity (e', m/s). The increase of this ratio is indicative of higher LV filling pressure.

OTHER OUTCOMES:
Change from baseline in Left Ventricular Stroke Volume after 12 months of treatment | March, 16th 2019 - March,16th 2020
  The LV stroke volume (in mL/beat) is obtained at echocardiography, as the product of the LV outflow tract area (cm2) and the time-velocity integral (cm) of the aortic flow velocity.
Change from baseline in Left Ventricular End-systolic Volume after 12 months of treatment | March, 16th 2019 - March,16th 2020
  The LV End-systolic volume (in mL) is calculated according to the biplane Simpson's method according to the recommendations of the American Society of Echocardiography and European Association of Cardiovascular Imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Frank L Dini, MD, Principal Investigator — Italian Society of Cardiology
Locations (1):
- Frank Lloyd Dini, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Metra M, Teerlink JR. Heart failure. Lancet. 2017 Oct 28;390(10106):1981-1995. doi: 10.1016/S0140-6736(17)31071-1. Epub 2017 Apr 28. PMID 28460827
- [Background] Januzzi JL Jr, Prescott MF, Butler J, Felker GM, Maisel AS, McCague K, Camacho A, Pina IL, Rocha RA, Shah AM, Williamson KM, Solomon SD; PROVE-HF Investigators. Association of Change in N-Terminal Pro-B-Type Natriuretic Peptide Following Initiation of Sacubitril-Valsartan Treatment With Cardiac Structure and Function in Patients With Heart Failure With Reduced Ejection Fraction. JAMA. 2019 Sep 17;322(11):1085-1095. doi: 10.1001/jama.2019.12821. PMID 31475295
- [Background] Mielniczuk LM, Tsang SW, Desai AS, Nohria A, Lewis EF, Fang JC, Baughman KL, Stevenson LW, Givertz MM. The association between high-dose diuretics and clinical stability in ambulatory chronic heart failure patients. J Card Fail. 2008 Jun;14(5):388-93. doi: 10.1016/j.cardfail.2008.01.015. Epub 2008 May 27. PMID 18514930
- [Background] Nohria A, Tsang SW, Fang JC, Lewis EF, Jarcho JA, Mudge GH, Stevenson LW. Clinical assessment identifies hemodynamic profiles that predict outcomes in patients admitted with heart failure. J Am Coll Cardiol. 2003 May 21;41(10):1797-804. doi: 10.1016/s0735-1097(03)00309-7. PMID 12767667
- [Background] Nagueh SF, Bhatt R, Vivo RP, Krim SR, Sarvari SI, Russell K, Edvardsen T, Smiseth OA, Estep JD. Echocardiographic evaluation of hemodynamics in patients with decompensated systolic heart failure. Circ Cardiovasc Imaging. 2011 May;4(3):220-7. doi: 10.1161/CIRCIMAGING.111.963496. Epub 2011 Mar 11. PMID 21398512
- [Background] Andersen OS, Smiseth OA, Dokainish H, Abudiab MM, Schutt RC, Kumar A, Sato K, Harb S, Gude E, Remme EW, Andreassen AK, Ha JW, Xu J, Klein AL, Nagueh SF. Estimating Left Ventricular Filling Pressure by Echocardiography. J Am Coll Cardiol. 2017 Apr 18;69(15):1937-1948. doi: 10.1016/j.jacc.2017.01.058. PMID 28408024
- [Background] Forrester JS, Diamond G, Chatterjee K, Swan HJ. Medical therapy of acute myocardial infarction by application of hemodynamic subsets (first of two parts). N Engl J Med. 1976 Dec 9;295(24):1356-62. doi: 10.1056/NEJM197612092952406. No abstract available. PMID 790191
- [Background] Stevenson LW, Perloff JK. The limited reliability of physical signs for estimating hemodynamics in chronic heart failure. JAMA. 1989 Feb 10;261(6):884-8. PMID 2913385
- [Background] Lechat P, Escolano S, Golmard JL, Lardoux H, Witchitz S, Henneman JA, Maisch B, Hetzel M, Jaillon P, Boissel JP, Mallet A. Prognostic value of bisoprolol-induced hemodynamic effects in heart failure during the Cardiac Insufficiency BIsoprolol Study (CIBIS). Circulation. 1997 Oct 7;96(7):2197-205. doi: 10.1161/01.cir.96.7.2197. PMID 9337190
- [Background] Hall SA, Cigarroa CG, Marcoux L, Risser RC, Grayburn PA, Eichhorn EJ. Time course of improvement in left ventricular function, mass and geometry in patients with congestive heart failure treated with beta-adrenergic blockade. J Am Coll Cardiol. 1995 Apr;25(5):1154-61. doi: 10.1016/0735-1097(94)00543-y. PMID 7897129
- [Background] Doughty RN, Whalley GA, Gamble G, MacMahon S, Sharpe N. Effects of carvedilol on left ventricular regional wall motion in patients with heart failure caused by ischemic heart disease. Australia-New Zealand Heart Failure Research Collaborative Group. J Card Fail. 2000 Mar;6(1):11-8. doi: 10.1016/s1071-9164(00)00007-5. PMID 10746814
- [Background] Konstam MA, Kronenberg MW, Rousseau MF, Udelson JE, Melin J, Stewart D, Dolan N, Edens TR, Ahn S, Kinan D, et al. Effects of the angiotensin converting enzyme inhibitor enalapril on the long-term progression of left ventricular dilatation in patients with asymptomatic systolic dysfunction. SOLVD (Studies of Left Ventricular Dysfunction) Investigators. Circulation. 1993 Nov;88(5 Pt 1):2277-83. doi: 10.1161/01.cir.88.5.2277. PMID 8222122
- [Background] Nicolosi GL, Latini R, Marino P, Maggioni AP, Barlera S, Franzosi MG, Geraci E, Santoro L, Tavazzi L, Tognoni G, Vecchio C, Volpi A. The prognostic value of predischarge quantitative two-dimensional echocardiographic measurements and the effects of early lisinopril treatment on left ventricular structure and function after acute myocardial infarction in the GISSI-3 Trial. Gruppo Italiano per lo Studio della Sopravvivenza nell'Infarto Miocardico. Eur Heart J. 1996 Nov;17(11):1646-56. doi: 10.1093/oxfordjournals.eurheartj.a014747. PMID 8922912
- [Background] Vardeny O, Claggett B, Kachadourian J, Desai AS, Packer M, Rouleau J, Zile MR, Swedberg K, Lefkowitz M, Shi V, McMurray JJV, Solomon SD. Reduced loop diuretic use in patients taking sacubitril/valsartan compared with enalapril: the PARADIGM-HF trial. Eur J Heart Fail. 2019 Mar;21(3):337-341. doi: 10.1002/ejhf.1402. Epub 2019 Feb 11. PMID 30741494
- [Background] Vardeny O, Claggett B, Kachadourian J, Pearson SM, Desai AS, Packer M, Rouleau J, Zile MR, Swedberg K, Lefkowitz M, Shi V, McMurray JJV, Solomon SD. Incidence, Predictors, and Outcomes Associated With Hypotensive Episodes Among Heart Failure Patients Receiving Sacubitril/Valsartan or Enalapril: The PARADIGM-HF Trial (Prospective Comparison of Angiotensin Receptor Neprilysin Inhibitor With Angiotensin-Converting Enzyme Inhibitor to Determine Impact on Global Mortality and Morbidity in Heart Failure). Circ Heart Fail. 2018 Apr;11(4):e004745. doi: 10.1161/CIRCHEARTFAILURE.117.004745. PMID 29643067
- [Background] McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, Rouleau JL, Shi VC, Solomon SD, Swedberg K, Zile MR; PARADIGM-HF Investigators and Committees. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014 Sep 11;371(11):993-1004. doi: 10.1056/NEJMoa1409077. Epub 2014 Aug 30. PMID 25176015
- [Background] Santos M, Rivero J, McCullough SD, West E, Opotowsky AR, Waxman AB, Systrom DM, Shah AM. E/e' Ratio in Patients With Unexplained Dyspnea: Lack of Accuracy in Estimating Left Ventricular Filling Pressure. Circ Heart Fail. 2015 Jul;8(4):749-56. doi: 10.1161/CIRCHEARTFAILURE.115.002161. Epub 2015 Jun 11. PMID 26067855
- [Background] Mullens W, Borowski AG, Curtin RJ, Thomas JD, Tang WH. Tissue Doppler imaging in the estimation of intracardiac filling pressure in decompensated patients with advanced systolic heart failure. Circulation. 2009 Jan 6;119(1):62-70. doi: 10.1161/CIRCULATIONAHA.108.779223. Epub 2008 Dec 15. PMID 19075104
- [Background] Nagueh SF. Non-invasive assessment of left ventricular filling pressure. Eur J Heart Fail. 2018 Jan;20(1):38-48. doi: 10.1002/ejhf.971. Epub 2017 Oct 8. PMID 28990316
- [Background] Dini FL, Ballo P, Badano L, Barbier P, Chella P, Conti U, De Tommasi SM, Galderisi M, Ghio S, Magagnini E, Pieroni A, Rossi A, Rusconi C, Temporelli PL. Validation of an echo-Doppler decision model to predict left ventricular filling pressure in patients with heart failure independently of ejection fraction. Eur J Echocardiogr. 2010 Sep;11(8):703-10. doi: 10.1093/ejechocard/jeq047. Epub 2010 Apr 17. PMID 20400763
- [Background] Farah E, Cogni AL, Minicucci MF, Azevedo PS, Okoshi K, Matsubara BB, Zanati SG, Haggeman R, Paiva SA, Zornoff LA. Prevalence and predictors of ventricular remodeling after anterior myocardial infarction in the era of modern medical therapy. Med Sci Monit. 2012 May;18(5):CR276-81. doi: 10.12659/msm.882732. PMID 22534706
- [Background] Gheorghiade M, Follath F, Ponikowski P, Barsuk JH, Blair JE, Cleland JG, Dickstein K, Drazner MH, Fonarow GC, Jaarsma T, Jondeau G, Sendon JL, Mebazaa A, Metra M, Nieminen M, Pang PS, Seferovic P, Stevenson LW, van Veldhuisen DJ, Zannad F, Anker SD, Rhodes A, McMurray JJ, Filippatos G; European Society of Cardiology; European Society of Intensive Care Medicine. Assessing and grading congestion in acute heart failure: a scientific statement from the acute heart failure committee of the heart failure association of the European Society of Cardiology and endorsed by the European Society of Intensive Care Medicine. Eur J Heart Fail. 2010 May;12(5):423-33. doi: 10.1093/eurjhf/hfq045. Epub 2010 Mar 30. PMID 20354029